CLINICAL TRIAL: NCT01659086
Title: An Observer-blind Study to Evaluate the Safety and Immunogenicity of GSK Biologicals' Influenza Vaccines GSK2654911A and GSK2654909A Administered to Adults 18 to 64 Years of Age
Brief Title: Study to Evaluate the Safety and Immunogenicity of GlaxoSmithKline (GSK) Biologicals' Influenza Vaccines GSK2654911A and GSK2654909A Administered to Adults 18 to 64 Years of Age
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 116358
Record Dates: First submitted 2012-08-03; First posted 2012-08-07 (Estimated); Last update posted 2018-06-18 (Actual); Status verified 2018-06

CONDITIONS: Influenza
Keywords: Influenza; Immunogenicity; H9N2; Safety
MeSH Terms: conditions — Influenza, Human

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor

ARMS (11):
- Group A (Experimental): Subjects will receive the investigational vaccine GSK2654911A formulation 1 and placebo
  Interventions: Biological: Investigational H9N2 vaccine GSK2654911A; Biological: Placebo
- Group B (Experimental): Subjects will receive the investigational vaccine GSK2654911A formulation 2 and placebo
  Interventions: Biological: Investigational H9N2 vaccine GSK2654911A; Biological: Placebo
- Group C (Experimental): Subjects will receive the investigational vaccine GSK2654911A formulation 3 and placebo
  Interventions: Biological: Investigational H9N2 vaccine GSK2654911A; Biological: Placebo
- Group D (Experimental): Subjects will receive the investigational vaccine GSK2654911A formulation 4 and placebo
  Interventions: Biological: Investigational H9N2 vaccine GSK2654911A; Biological: Placebo
- Group E (Experimental): Subjects will receive the investigational vaccine GSK2654909A and placebo
  Interventions: Biological: Investigational H9N2 vaccine GSK2654909A; Biological: Placebo
- Group F (Experimental): Subjects will receive the investigational vaccine GSK2654911A formulation 5
  Interventions: Biological: Investigational H9N2 vaccine GSK2654911A
- Group G (Experimental): Subjects will receive the investigational vaccine GSK2654911A formulation 6
  Interventions: Biological: Investigational H9N2 vaccine GSK2654911A
- Group H (Experimental): Subjects will receive the investigational vaccine GSK2654911A formulation 7
  Interventions: Biological: Investigational H9N2 vaccine GSK2654911A
- Group I (Experimental): Subjects will receive the investigational vaccine GSK2654911A formulation 8
  Interventions: Biological: Investigational H9N2 vaccine GSK2654911A
- Group J (Experimental): Subjects will receive the investigational vaccine GSK2654909A
  Interventions: Biological: Investigational H9N2 vaccine GSK2654909A
- Placebo Group (Placebo Comparator): Subjects will receive Placebo
  Interventions: Biological: Placebo

INTERVENTIONS:
Biological: Investigational H9N2 vaccine GSK2654911A — 2 or 3 doses of GSK2654911A (different formulations) followed by 1 or 0 dose of saline placebo respectively, depending in the treatment group. All doses to be administered intramuscularly (IM) in deltoid region of arm.
  Arms: Group A; Group B; Group C; Group D; Group F; Group G; Group H; Group I
Biological: Investigational H9N2 vaccine GSK2654909A — 2 or 3 doses of GSK2654909A followed by 1 or 0 dose of saline placebo, respectively (treatment 5). All doses to be administered IM in deltoid region of arm.
  Arms: Group E; Group J
Biological: Placebo — 1 dose of saline placebo administered intramuscularly (IM) in deltoid region of arm.
  Arms: Group A; Group B; Group C; Group D; Group E; Placebo Group

SUMMARY:
The purpose of this study is to evaluate the safety, reactogenicity, and immunogenicity of different formulations of a two-dose primary series and booster vaccination of monovalent Influenza H9N2 vaccine manufactured in Quebec, Canada with and without adjuvant, in adults 18 to 64 years of age.

ELIGIBILITY:
Inclusion Criteria:

* Male or female adults from 18 to 64 years of age (inclusive) at time of first study vaccination.
* Written informed consent obtained from the subject.
* Subjects who the investigator believes can and will comply with the requirements of the protocol.
* Healthy subjects as established by medical history and physical examination.
* Body weight of at least 110 lbs (49.9 kg).
* Access to a consistent means of telephone contact, which may be either in the home or at the workplace, land line or mobile, but NOT a pay phone or other multiple-user device (i.e., a common-use phone serving multiple rooms or apartments).
* Female subjects of non-childbearing potential may be enrolled in the study. Non-childbearing potential is defined as current tubal ligation, hysterectomy, ovariectomy or post-menopause.
* Female subjects of childbearing potential may be enrolled in the study, if they have practiced adequate contraception for 30 days prior to vaccination, and have a negative pregnancy test on the day of vaccination, and agree to continue to practice adequate contraception until 2 months after booster dose administration.

Exclusion Criteria:

* Presence or evidence of neurological or psychiatric diagnoses which, although stable, are deemed by the investigator to render the potential subject unable/unlikely to provide accurate safety reports.
* Presence or evidence of substance abuse.
* Diagnosed with cancer, or treatment for cancer within three years.

  * Persons with a history of cancer who are disease-free without treatment for three years or more are eligible.
  * Persons with a history of histologically-confirmed basal cell carcinoma of the skin successfully treated with local excision only are excepted and may enroll, but other histologic types of skin cancer are exclusionary.
  * Women who are disease-free three years or more after treatment for breast cancer and receiving long-term prophylaxis may enroll.
* Presence of a temperature ≥ 38.0ºC (≥100.4ºF), or acute symptoms greater than "mild" severity on the scheduled date of first vaccination.
* Any confirmed or suspected immunosuppressive or immunodeficient condition including history of human immunodeficiency virus (HIV) infection (no laboratory testing required).
* Receipt of systemic glucocorticoids (e.g., prednisone ≥ 10 mg/day for more than 14 consecutive days) within 30 days prior to the first dose of study vaccine, or any other cytotoxic, immunosuppressive or immune-modifying drugs within 365 days of study enrollment. Topical, intra-articularly injected, or inhaled glucocorticoids, topical calcineurin inhibitors or imiquimod are allowed.
* Any significant disorder of coagulation or treatment with warfarin derivatives or heparin. Persons receiving individual doses of low molecular weight heparin outside of 24 hours prior to vaccination are eligible. Persons receiving prophylactic antiplatelet medications, e.g., low-dose aspirin, and without a clinically-apparent bleeding tendency, are eligible.
* An acute evolving neurological disorder or Guillain Barré Syndrome within 42 days of receipt of prior seasonal or pandemic influenza vaccine.
* Administration of an inactive vaccine within 14 days or of a live attenuated vaccine within 30 days before the first dose of study vaccine/product.
* Planned administration of any vaccine other than the study vaccine/product before blood sampling at the Day 42 visit.
* Previous administration of any H9 vaccine or physician-confirmed H9 disease.
* Use of any investigational or non-registered product other than the study vaccine within 30 days preceding the first dose of study vaccine, or planned use during the study period.
* Receipt of any immunoglobulins and/or any blood products within 90 days before study enrolment or planned administration of any of these products during the study period.
* Any known or suspected allergy to any constituent of influenza vaccines or component used in the manufacturing process of the study vaccine including a history of anaphylactic-type reaction to consumption of eggs; or a history of severe adverse reaction to a previous influenza vaccine.
* Known pregnancy or a positive urine beta-human chorionic gonadotropin (β-hCG) test result before the first vaccination.
* Lactating or nursing women.
* Any condition which, in the opinion of the investigator, prevents the subject from participating in the study.

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 422 (Actual)
Dates: Start 2012-08-22 (Actual); Primary Completion 2012-10-26 (Actual); Study Completion 2014-03-19 (Actual)

PRIMARY OUTCOMES:
Humoral immune response in terms of HI antibodies against H9N2 v-like antigen | Day 21
Humoral immune response in terms of HI antibodies against H9N2 v-like antigen | Day 42

SECONDARY OUTCOMES:
Humoral immune response in terms of HI antibodies against H9N2 antigen | GMTs and seropositivity rates, SPR on Days 0, 7, 21, 28, 42, 182, 191, 385 and 546. SCR and MGI on Days 7, 21, 28, 42, 182, 191, 385 and 546. B-SCR and BF on Days 191, 385 and 546.
Humoral immune response in terms of HI antibodies against H9N2 antigen for each vaccine group and for age strata (18-40 years; 41-64 years) | GMTs and seropositivity rates, SPR on Days 0, 7, 21, 28, 42, 182, 191, 385 and 546. SCR and MGI on Days 7, 21, 28, 42, 182, 191, 385 and 546. B-SCR and BF on Days 191, 385 and 546.
Humoral immune response in terms of HI antibodies against any drift strain from H9N2 antigen or against any other H9 subtype antigen | GMTs and seropositivity rates on Days 0, 7, 21, 28, 42, 182 , 191, 385 and 546. SCR and MGI on Days 21, 42, 182, 191, 385, 546. SPR on Days 0, 21, 42, 182, 191, 385 and 546. B-SCR and BF on Days 191, 385 and 546.
Humoral immune response in terms of neutralizing (MN) antibodies against H9N2 and against any drift strain (or other H9 subtype) | GMTs and seropositivity rate on Days 0, 21, 42, 182, 191, 385 and 546. VRR on Days 21, 42, 182, 191, 385, 546. Booster-VRR on Day 191, 385 and 546.
Occurrence of local and general symptoms | During the 7-day follow-up period (i.e., day of vaccination and 6 subsequent days) after any vaccination
Occurrence and relationship to vaccination of unsolicited adverse events | Within 21 days (Day 0 to Day 20, 21 to 41, 182 to 202) after any vaccination
Occurrence and relationship to vaccination of adverse events with medically attended visits | During the entire study period (Day 0 - Day 546)
Occurrence and relationship to vaccination of Adverse events of special interest (AESIs), potential Immune-Mediated Diseases (pIMDs), Serious Adverse Events (SAEs) and adverse pregnancy outcome | During the entire study period (Day 0 - Day 546)
Number of subjects with clinical safety laboratory abnormalities | Days 0, 7, 21, 28, 42, 182, 191, and 385.

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (4):
- United States (3):
  - GSK Investigational Site, Miami, Florida
  - GSK Investigational Site, Edison, New Jersey
  - GSK Investigational Site, Austin, Texas
- GSK Investigational Site, Sherbrooke, Quebec, Canada

IPD SHARING:
Plan to Share IPD: Yes
IPD for this study will be made available via the Clinical Study Data Request site.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: IPD is available via the Clinical Study Data Request site (click on the link provided below)
Access Criteria: Access is provided after a research proposal is submitted and has received approval from the Independent Review Panel and after a Data Sharing Agreement is in place. Access is provided for an initial period of 12 months but an extension can be granted, when justified, for up to another 12 months.
URL: https://clinicalstudydatarequest.com

REFERENCES:
- [Derived] Madan A, Collins H, Sheldon E, Frenette L, Chu L, Friel D, Drame M, Vaughn DW, Innis BL, Schuind A. Evaluation of a primary course of H9N2 vaccine with or without AS03 adjuvant in adults: A phase I/II randomized trial. Vaccine. 2017 Aug 16;35(35 Pt B):4621-4628. doi: 10.1016/j.vaccine.2017.07.013. Epub 2017 Jul 15. PMID 28720281
- See also: Results for study 116358 can be found on the GSK Clinical Study Register — https://www.gsk-clinicalstudyregister.com/study/116358?search=study&b%22b''%22#rs